CLINICAL TRIAL: NCT02568995
Title: Postoperative Pain Management Following Total Hip Arthroplasty. A Comparison Between Local Infiltration Analgesia and Ultrasound Guided 3-in-1 Block
Brief Title: Pain Management Following Total Hip Arthroplasty
Acronym: FEMORALIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Anil Gupta, Associate Professor, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THA2014
Record Dates: First submitted 2015-10-02; First posted 2015-10-06 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Postoperative Pain Intensity; Rescue Pain Requirements
Keywords: postoperative pain; morphine; total hip arthroplasty; femoral nerve block
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Ketorolac; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LIA (Experimental): Local infiltration analgesia using a combination of ropivacaine 300 mg + ketorolac 30 mg + adrenaline 0.5 mg
  Interventions: Drug: ropivacaine + ketorolac + adrenaline
- Femoral nerve block (Active Comparator): Ultrasound guided 3-in-1 block using 30 ml of 0.75% ropivacaine
  Interventions: Drug: ropivacaine + ketorolac + adrenaline

INTERVENTIONS:
Drug: ropivacaine + ketorolac + adrenaline — A combination of drugs injected locally for postoperative pain management

SUMMARY:
Total hip arthroplasty (THA) is a common and standardized procedure. Postoperative mortality after hip joint replacement is low but some complications remain, including chronic post-surgical pain (1), hip dislocation (2), infection (3), and deep vein thrombosis (4). Strategies that have been identified to reduce morbidity and mortality include: posterior surgical approach, mechanical and pharmacological prophylaxis of deep vein thrombosis, and the use of spinal anesthesia (5). One of the important factors for patient satisfaction with lower limb arthroplasty is good postoperative pain management (6). Poorly managed postoperative pain can lead to chronic post-surgical pain and therefore aggressive postoperative pain management is important (7). Several different methods have been used to treat postoperative pain following THA. Recently, local infiltration analgesia (LIA) using a combination of large volume local anesthetics (LA) and non-steroidal anti-inflammatory agents (NSAID) injected systematically peri-articularly has been used for pain management with variable success (8). We found that better analgesia could be achieved when using LIA compared to intrathecal morphine during the first few days postoperatively (9,10).

Ultrasound techniques are commonly used for peripheral nerve blocks and have been shown to reduce pain intensity and may be considered by many to be a standard of care. Specifically, the 3-in-1 block has been commonly used because of its ease of application and good pain management following total hip arthroplasty. The present study aims to compare postoperative pain intensity following local infiltration analgesia with a standardised 3-in-1 block for total hip arthroplasty.

DETAILED DESCRIPTION:
Sixty ASA I-II patients undergoing THA would be randomised to one of two groups in a double-blind study:

Group LIA: A total of 151.5 ml of a combination of 0.2% ropivacaine (150 ml), 30 mg ketorolac (1 ml) and 0.5 mg (0.5 ml) adrenaline was administered systematically peri-articularly during THA and 30 ml of normal saline for ultrasound-guided 3-in-1 block Group Femoral block: Received 30 ml of ropivacaine 0,75% for ultrasound-guided 3-in-1 block and a total of 151.5 ml of normal saline peri-articularly.

All patients would receive spinal anaesthesia with 0.5% heavy bupivacaine for surgery

Postoperatively, the following parameters would be measured:

1. Pain intensity at fixed time intervals during 0-7 days and thereafter at weekly intervals for 1 month
2. Rescue morphine consumption during 0-4, 4-24 and 24-48 h
3. Side effects and complications
4. Home readiness and length of hospital stay
5. Chronic pain intensity measured after 3 and 6 months using the Brief Pain Inventory
6. Plasma Cytokine concentration at fixed intervals
7. Motor block using Bromage scale
8. EQ5D and HOOS questionnaires

ELIGIBILITY:
Inclusion Criteria:

* 40-80 years
* ASA I-II
* THA operation

Exclusion Criteria:

* Chronic pain requiring opiates
* Language constraints preventing completion of the study
* Contraindications to regional block

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 24 h
  Pain intensity during movement at 24 h after end of surgery

SECONDARY OUTCOMES:
Rescue analgesic consumption | 0-24 h
  Amount of PCA morphine used for pain management
Chronic pain | 3-6 months
  Pain at 3 and 6 months after surgery using Brief Pain Inventory
Inflammation | Preoperative to 3-5 days postoperatively
  Pre- and post-operative cytokine concentration would be measured

CONTACTS AND LOCATIONS:
Locations (3):
- Sweden (3):
  - University Hospital, Örebro
  - Örebro University Hospital, Örebro
  - Karolinskasjukhuset, Solna